CLINICAL TRIAL: NCT01872949
Title: C-Pulse System eurOPean mulTicenter Study, Implantable cOuNterpulsation System in patIents With Moderate to Severe Heart Failure
Brief Title: C-Pulse® System European Multicenter Study
Acronym: OPTIONS-HF
Status: Completed | Type: Observational
Sponsor: Nuwellis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO 04654-C
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; NYHA Class III; NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to observe the clinical outcomes of heart failure patients treated with C-Pulse® System in the usual manner and according to the approved indications and contraindications.

DETAILED DESCRIPTION:
Evaluation of the post-market clinical performance and safety of the C-Pulse® System for the treatment of Heart Failure in the population of patients who meet the approved clinical conditions provided in the indications and contraindications.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older
* Patients with moderate to severe ambulatory heart failure [American College of Cardiology/American Heart Association (ACC/AHA) Stage C; NYHA Class III/IV ambulatory], who are refractory to optimal medical therapy
* Patients who are non-responders to CRT pacemaker therapy
* Patient has signed and dated the investigation informed consent form

Exclusion Criteria:

* Evidence of significant ascending aortic calcification on postero-anterior chest X-ray or CT scan
* Moderate or severe atherosclerotic aortic disease
* Ascending aorto-coronary artery bypass grafts
* Any history of aortic dissection
* Connective tissue disorder such as Marfans disease
* Aorta not conforming to specified dimensional constraints
* Patient has severe mitral valve incompetence, grade 4+
* Patient has moderate to severe aortic valve incompetence, grade 2 - 4+
* Patient has systolic blood pressure less than 90 or greater than 140mmHg
* Presence of active systemic infection
* Presence of bleeding or coagulation disorder (relative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient population of up to 50 patients with moderate to severe heart failure refractory to optimal medical therapy, who are implanted with the C-Pulse System as clinically appropriate, will be enrolled into the Study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- University Hospital, Innsbruck, Austria
- Germany (7):
  - Evangelisches Krankenhaus Niederrhein, Duisburg, Northrhine-Westfalia
  - Cardio-Centrum Berlin, Berlin
  - Vivantes Klinikum, Berlin
  - Unfallkrankenhaus, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Medizinische Hochschule, Hanover
  - Universität Tübingen, Tübingen

REFERENCES:
- [Derived] Schulz A, Krabatsch T, Schmitto JD, Hetzer R, Seidel M, Dohmen PM, Hotz H. Preliminary Results From the C-Pulse OPTIONS HF European Multicenter Post-Market Study. Med Sci Monit Basic Res. 2016 Feb 18;22:14-9. doi: 10.12659/MSMBR.896959. PMID 26887528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The OPTIONS-HF is a prospective, post-market, open label study designed to enroll up to 50 patients in up to fifteen (15) European sites. Only 15 subjects were implanted.
Groups:
- C-Pulse System: Single-arm study
Period: Overall Study
Arm/Group | C-Pulse System
Started | 15
Completed | 4
Not Completed | 11

BASELINE CHARACTERISTICS:
Units Other Than Participants: implants
Groups:
- C-Pulse System: A total of 15 subjects were treated with the C-Pulse System.
Arm/Group | C-Pulse System
Number analyzed (Participants) | 15
Number analyzed (implants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9.3)
Age, Customized [Median (Full Range); unit: years]
  Median | 61 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: European Caucasian | 14
  Race: Subject Choose not to Provide | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1
  Germany | 13
  United Kingdom | 1
NYHA Classification [Count of Participants; unit: Participants] — NYHA Classification provides a simple way of classifying the extent of heart failure.
  Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    I | 0
    II | 0
    III | 14
    IV | 1
INTERMACS Subject Profile/Status [Count of Participants; unit: Participants] — 1. Critical Cardiogenic Shock, 2. Progressive Decline, 3. Stable but Inotrope Dependent, 4. Resting Symptoms, 5. Exertion Intolerant, 6. Exertion Limited, 7. Advanced NYHA Class III, or 8. NA/NYHA class I or II
  Participants
    Resting Symptoms | 3
    Exertion Intolerant | 5
    Exertion Limited | 4
    Advanced NYHA Class III | 1
    NA, NYHA class I or II | 2
Six Minute Walk Test [Mean (Standard Deviation); unit: meters] — The six minute walk test (6MWT) is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. Walking is an activity performed daily by all but the most severely impaired patients. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD).
  meters | 237.4 (85.6)
Kansas City Cardiomyopathy Questionnaire [Mean (Standard Deviation); unit: points] — The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. Population: Number analyzed is different from overall participants because one participant did not take the KCCQ.
  points
    number analyzed (Participants) | 14
    (all) | 30 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Survival and Study Completion
Description: Amount of participants that did not exit study for reasons including worsening heart failure resulting in hospitalization, LVAD implantation, study withdrawal or death.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | C-Pulse System
Number analyzed (Participants) | 15
Participants
  Exited Study | 11
  Study completion | 4

2. Primary Outcome: NYHA Classification
Description: Participant NYHA Classification at 6 month follow up. The NYHA Classification involved 4 classes.
  I No limitation of physical activity II Slight limitation of physical activity III Marked limitation of physical activity IV Unable to carry on any physical activity without discomfort
Time Frame: 6 Months
Population: Only 12 participants remained in the study at the 6-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | C-Pulse System
Number analyzed (Participants) | 12
Participants
  NYHA Class I | 2
  NYHA Class II | 6
  NYHA Class III | 4
  NYHA Class IV | 0

3. Primary Outcome: INTERMACS Subject Profile/Status
Description: 1. Critical Cardiogenic Shock, 2. Progressive Decline, 3. Stable but Inotrope Dependent, 4. Resting Symptoms, 5. Exertion Intolerant, 6. Exertion Limited, 7. Advanced NYHA Class III, 8. NA/NYHA class I or II
Time Frame: 6 months
Population: Only 12 participants remained in the study at the 6-Month follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- C-Pulse System: A total of 15 subjects were treated with the C-Pulse System. The study follow-up period was up to 5 years. However, the data collection for subjects was up to 24-months. Only 3 subjects completed the 24 months follow-up visit, and 12 subjects prematurely exited the study prior to the 24 months follow-up.
Arm/Group | C-Pulse System
Number analyzed (Participants) | 12
Participants
  Resting Symptoms | 1
  Exertion Limited | 1
  Advanced NYHA Class III | 2
  NA, NYHA class I or II | 8

4. Primary Outcome: Six Minute Walk Test
Description: The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Time Frame: 6 months
Population: Only 9 participants were able to be assessed via 6MWT at the 6-Month follow-up.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | C-Pulse System
Number analyzed (Participants) | 9
Meters | 333.9 (112.2)

5. Primary Outcome: KCCQ
Description: Overall score from Kansas City Cardiomyopathy Questionnaire, a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status,which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. Scores range from 0-100, in which higher scores reflect better health status.
Time Frame: 6 months
Population: Only 12 participants were involved in the study at the time of KCCQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Pulse System
Number analyzed (Participants) | 12
score on a scale | 60.3 (21.1)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Events for the C-Pulse European study were reported by Investigators using the INTERMACS ™ Adverse Event Definitions as a guideline.
Groups:
- C-Pulse System: A total of 15 subjects were treated with the C-Pulse System. The study follow-up period was up to 5 years. However, the data collection for subjects was up to 24-months. Only 3 subjects completed the 24 months follow-up visit, and 12 subjects prematurely exited the study prior to the 24 months follow-up. \Rate subjects with averse event 93% (14/15).
Arm/Group | C-Pulse System
All-Cause Mortality (participants affected / at risk) | 6/15
Serious Adverse Events (participants affected / at risk) | 14/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C-Pulse System (N=15)
Major Infection (Infections and infestations) | 7 (8) — A clinical infection accompanied by pain, fever, drainage and/or leukocytosis that is treated by anti-microbial agents (non-prophylactic).
Cardiac Arrhythmias (Cardiac disorders) | 5 (5) — Including sustained ventricular and supraventricular arrhythmias
Worsening Left Heart Failure (Cardiac disorders) | 5 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C-Pulse System (N=15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT01872949/Prot_SAP_000.pdf